CLINICAL TRIAL: NCT01037569
Title: Optimizing Toxicological Screening in Drug Endangered Children
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907431; 07-DA-N431
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-22

CONDITIONS: Substance Abuse Detection
Keywords: Toxicological Screening; Drugs; Alternative Matrices; Urine; Children

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Children who enter the foster care system are all too often exposed to illicit drugs in the home. Children from these homes, known as drug endangered children, are not routinely tested for harmful substances. Any short- and long-term physical or developmental problems they may experience as a result of this exposure often go undetected and untreated.
* Children who are placed into protective custody are not always screened by physicians or nurse practitioners. Although drug-endangered children under 18 years of age automatically receive a urine toxicology screen to determine the types and levels of illicit drugs in their systems, this procedure has difficulties and limitations that may affect the quality of the data. Researchers are interested in developing more effective methods of analyzing the presence or absence of illicit environmental drug exposure in children.

Objectives:

- To determine the most effective method of identifying long-term illicit stimulant drug exposure in drug-endangered children.

Eligibility:

- Children under 18 years of age who are being placed into protective custody after having been found in a home where drugs are manufactured, used, or sold.

Design:

* Researchers will gain verbal consent for the procedure for children who are 7 years of age or older. Children younger than 7 years of age will not be required to give verbal consent for sample collection.
* Researchers will collect standard urine samples for toxicological screening. Part of the sample will be sent to the National Institute on Drug Abuse for evaluation; the rest will remain with the local authority.
* In addition to this standard procedure, researchers will collect a hair sample by cutting a small amount of hair from the crown of the head as close to the root as possible (and not pulling any hair out of the child's head).
* Researchers will also use an oral swab to collect a saliva sample from the inside cheek of each child.
* No clinical care will be provided under this protocol....

DETAILED DESCRIPTION:
This is a single-center, investigator-initiated study to determine the best method for analyzing the presence or absence of illicit environmental drug exposure in children placed into protective custody in Sacramento County. In collaboration with the National Institutes of Health (NIH), National Institute of Drug Abuse (NIDA) we will use diagnostic procedures to determine the presence of illicit drugs in the following three samples: (1) hair; (2) oral swab; and (3) urine. These samples will be sent to a designated NIH lab site where 100 de-identified samples will be analyzed for methamphetamine, amphetamine, Ecstasy (MDMA), and MDEA.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Inclusion criteria are the following (and must have all of the following):

1. children under the age of 18 (the vast majority - 87 percent - of children examined at the Center are under the age of 6);
2. children placed into protective custody by Sacramento County CPS or law enforcement;
3. children examined at the CAARE Center; and
4. children found in a home where drugs are manufactured, used and/or sold.

Exclusion criteria are the following (any one of the following may apply):

1. anyone who has reached the age of majority;
2. those found to have parents who are not drug abusers;
3. those where there was no definitive evidence of environmental drug exposure (i.e., suspicious parent, but no drugs were found in the home); or
4. any child, drug exposed or not, who is examined in the UCD Emergency Department (after hours - 9:00 pm to 7:00 am - and weekends).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07-10; Study Completion 2011-03-22

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States